## Statistical Analysis Plan

Clinical trial protocol title: A microdose Study to Evaluate the Biodistribution of

[<sup>11</sup>C]-GSK2256098 in the Lungs and Heart of Healthy Subjects and Pulmonary Arterial Hypertension (PAH) Patients using Positron Emission Tomography (PET)

HMR code: 15-505

EudraCT no: 2015-002626-40

CRO details: Hammersmith Medicines Research

Cumberland Avenue London NW10 7EW

Sponsor details: GlaxoSmithKline Research & Development Limited

980 Great West Road

Brentford

Middlesex, TW8 9GS

UK

Issued: 4 October 2016

Version: 1.1

Based on: Protocol Amendment 03, 22 April 2016

Number of pages: 46

Prepared by:

## **Table of contents**

| LIST | OF ABBREVIATIONS | 4 |
|---|---|---|
| SIGN | NATURES | 5 |
| INTE | RODUCTION | 6 |
| STUI | DY OBJECTIVE(S) AND ENDPOINT(S) | 6 |
| 4.1 | Study Objective(s) | 6 |
| | 4.1.1 Primary Objective(s) | 6 |
| | 4.1.2 Exploratory Objective(s) | 6 |
| 4.2 | Study Endpoint(s) | 7 |
| | 4.2.1 Primary Endpoint(s) | 7 |
| | 4.2.2 Exploratory Endpoint(s) | 7 |
| 4.3 | Statistical Hypotheses | 7 |
| TIMI | E AND EVENTS TABLE | 8 |
| PLA | NNED ANALYSES | 10 |
| 7.1 | Interim Analyses | 10 |
| | 7.1.1 Persons responsible for analysis | 10 |
| 7.2 | • | |
| SAM | | |
| 8.1 | Sample Size Re-estimation or Adjustment | 11 |
| ANA | LYSIS POPULATIONS | 12 |
| 9.1 | Analysis Datasets | 12 |
| TRE | ATMENT COMPARISONS | 12 |
| GEN | ERAL CONSIDERATIONS FOR DATA ANALYSES | 12 |
| 11.1 | Data Display Group Descriptors | 12 |
| 11.2 | Conventions for Summary Statistics and Data Displays | 13 |
| DAT | A HANDLING CONVENTIONS | 13 |
| 12.1 | Premature Withdrawal and Missing Data | 13 |
| 12.2 | Derived and Transformed Data | 13 |
| 12.3 | Assessment Windows | 14 |
| 12.4 | Values of Potential Clinical Importance | 14 |
| STUI | DY POPULATION | 14 |
| 13.1 | Disposition of Subjects | 14 |
| 13.2 | Protocol Deviations | 15 |
| | SIGN INTE STUI 4.1 4.2 4.3 STUI TIMI PLAI 7.1 7.2 SAM 8.1 ANA 9.1 TRE GEN 11.1 11.2 DAT 12.1 12.2 12.3 12.4 STUI 13.1 | 4.1.1 Primary Objective(s) 4.1.2 Exploratory Objective(s) 4.2.1 Primary Endpoint(s) 4.2.1 Primary Endpoint(s) 4.2.2 Exploratory Endpoint(s) 4.3 Statistical Hypotheses STUDY DESIGN |

| | 13.3 | Demographic and Baseline Characteristics | 15 |
|-----|--------|---------------------------------------------------|----|
| | 13.4 | Treatment Compliance | 16 |
| 14 | SAFE | ETY ANALYSES | 16 |
| | 14.1 | Adverse Events | 16 |
| | 14.2 | Deaths, Cardiovascular and Serious Adverse Events | 16 |
| | 14.3 | Other Safety Measures | 17 |
| | | 14.3.1 Clinical Laboratory Evaluations | 17 |
| | | 14.3.2 Vital signs | 17 |
| | | 14.3.3 Physical examination | 17 |
| | 14.4 | Positron Emission Tomography | 17 |
| 15 | REFI | ERENCES | 19 |
| 16 | ATT | ACHMENTS | 19 |
| | 16.1 | Data Display Requirements | 19 |
| | 16.2 | Table of Contents for Data Display Specifications | 20 |
| | 16.3 | Data Display Specifications | 24 |
| | | 16.3.1 Table Outlines | 24 |
| | | 16.3.2 Figure Outlines | 33 |
| | | 16.3.3 Listing Outlines | 35 |
| APP | PENDIX | A: LABORATORY RANGES | 44 |
| APP | PENDIX | B: SAMPLE PAGE LAYOUT | 46 |

## 1 List of abbreviations

| AΕ | Adverse Event |
|--------|----------------------------------------------|
| APTT | Activated Partial Thromboplastin Time |
| BMI | Body Mass Index |
| CRF | Case Report Form |
| CT | Computerised Tomography |
| CTR | Clinical Trial Report |
| ECG | Electrocardiogram |
| FAK | Focal adhesion kinase |
| GSK | GlaxoSmithKline |
| HIV | Human Immunodeficiency Virus |
| HMR | Hammersmith Medicines Research |
| HPD | Highest Posterior Density |
| | - |
| HV | Healthy Volunteers |
| ICH | International Conference on Harmonization |
| IMP | Investigational Medicine Product |
| INR | International Normalised Ratio |
| IPF | Idiopathic Pulmonary Fibrosis |
| MCMC | Monte Carlo Markov Chain |
| MedDRA | Medical Dictionary for Regulatory Activities |
| N | Number of subjects |
| n | Number of observed subjects |
| PAH | Pulmonary Arterial Hypertension |
| PDF | Portable Document Format |
| PET | Positron Emission Tomography |
| PT | Prothrombin Time |
| Q1 | Lower quartile |
| Q3 | Upper quartile |
| ROI | Region of Interest |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SD | Standard deviation |
| SUV | Standardised Uptake Value |
| TEAE | Treatment-Emergent Adverse Event |
| TT | Thrombin time |
| T/T | |
| VT | Volume of Distribution |

## 2 Signatures

The following persons have read and agreed the content of this Statistical Analysis Plan:



#### 3 Introduction

This Statistical Analysis Plan (SAP) is based on the current trial protocol (Amendment 3, 22Apr2016) and CRF (version 1, 28Sep2015). Where statistical methods differ substantially between this SAP and the protocol, that will be identified in this document.

This SAP describes the datasets and the statistical methods to be used for the reporting and analysis of all data collected during the trial except then genetics sample data.

If a future protocol amendment necessitates a substantial change to the statistical analysis of the trial data, this SAP will be amended accordingly. If, after database lock, additional analyses are required to supplement the planned analyses described in this SAP, those unplanned analyses will not be described in an amended SAP, but they will be identified in the integrated clinical trial report (CTR). Any deviations from this SAP will be documented in the CTR.

This SAP has been written in consideration of the following guidelines:

- International Conference on Harmonization (ICH) E9, Guidance for Industry: Statistical Principles for Clinical Trials (ICH E9 1998)1; and
- ICH E3, Guidance for Industry: Structure and Content of Clinical Study Reports (ICH E3 1995)2.

Statistical analysis will be done using SAS® 9.3 on a Windows PC.

## 4 Study Objective(s) and Endpoint(s)

## 4.1 Study Objective(s)

#### 4.1.1 Primary Objective(s)

To compare the uptake of [11C]-GSK2256098 in the heart and lungs of PAH patients versus the heart and lungs of healthy control subjects

#### 4.1.2 Exploratory Objective(s)

To explore the spatial distribution of [<sup>11</sup>C]-GSK2256098 uptake in the heart and lungs of PAH patients versus the heart and lungs of healthy control subjects.

## 4.2 Study Endpoint(s)

### 4.2.1 Primary Endpoint(s)

Uptake of [ $^{11}$ C]-GSK2256098 in the heart and lung (assessed as the volume of distribution ( $V_T$ ) and/or standardised uptake values (SUV)) as measured by PET

### 4.2.2 Exploratory Endpoint(s)

Qualitative assessment of the spatial distribution of [11C]-GSK2256098 uptake in the heart and lungs

### 4.3 Statistical Hypotheses

No formal statistical testing will be done. Instead an estimation approach has been adopted. Simple Bayesian methods will be used to quantify the evidence which the study generates about the endpoints themselves, and about contrasts (probability ratios) of these endpoints.

## 5 Study Design

This is cross-sectional study exploring the uptake of [<sup>11</sup>C]-GSK2256098 in PAH patients and in healthy (age and gender-matched) volunteers.

It is a non-randomised, open label study where all volunteers will receive one microdose of the radiolabelled compound.

Up to 12 healthy subjects and 12 PAH patients (including those with a prolonged QTcF interval  $\leq$  500ms) will be enrolled to provide sufficient PET data to quantify the uptake of [11C]-GSK2256098 in the heart and lungs.

## **6** Time and Events Table

| Procedure | Screening (up to 30 days prior to scan) | Scanning visit | Follow-up (2-4 weeks post-last dose) | Notes |
|---|---|---|---|---|
| Informed consent | X | | | |
| Inclusion and exclusion criteria | X | | | |
| Demography | X | | | |
| Brief physical | х | X | X | On the scanning day, to be completed pre-scan, prior to the administration of the peptide. |
| Medical / Medical history | X | | | |
| Vital signs | X | X | | On the scanning day, to be conducted pre and post scan. |
| 12-lead ECG | X | | | |
| Alcohol breath test | X | X | | |
| Urine drug and cotinine screen | X | | | |
| Healthy subjects only: spirometry | X | | | |
| Coagulation profile | X | | | This will include PT (Prothrombin time), APTT (Activated Partial Thromboplastin Time) and Thrombin Time (TT) |
| PAH patients only (who have been on<br>Warfarin): INR | | X | | Sample to confirm suitability for scanning day can be done up to 3 days prior to the day of the scan |
| HIV, Hep B and Hep C screen | X | | | If test otherwise performed within 3 months prior to<br>first dose of study treatment, testing at screening is<br>not required |
| Clinical chemistry and Haematology | X | | | |
| Urinalysis | X | | | |
| Allen's test | X | X | | |
| i.v dose of [11C]-GSK2256098 | | X | | |
| PET scan | | X | | PET scanning will be started at the same time as injection of the radioligand and PET data will be collected for up to 90 minutes post administration. |

| Procedure | Screening (up to 30 days prior to scan) | Scanning visit | Follow-up (2-4 weeks post-last dose) | Notes |
|---|---|---|---|---|
| Attenuation CT scan | | X | | Lasting seconds to minute prior to start of PET scan. If subject gets off the bed for a comfort break midway through the PET scan, another CT scan will be performed prior to re-starting acquisition of PET data |
| Genetics sample | | X | | Genetic Informed consent must be obtained before collecting a sample |
| Samples for plasma radioactivity measurements & whole blood | | X | | Blood samples will be collected during scanning for plasma and whole blood radioactivity measurements. |
| AE/SAE review | | X | X | |
| Concomitant medication review | X | X | X | |

## 7 Planned Analyses

## 7.1 Interim Analyses

No formal interim "testing" of any statistical hypothesis will be performed.

The strength of evidence in the PET data (about differential expression levels between patients and HVs) will be reviewed once five patients and five healthy volunteers have been studied in the PET scanner, and the relevant functional endpoints have been derived by Imanova scientists for heart chamber and whole lung regions. From that point onwards, the data will be monitored continuously (or as near as possible given practicalities of study operationalisation)

#### 7.1.1 Persons responsible for analysis



## 7.2 Final Analysis

The database will be locked once all subjects have completed the study, data have been entered and all queries resolved. The final analysis will be carried out following database lock.

#### 7.2.1 Persons responsible for analysis



## 8 Sample Size Considerations

There is little known about the likely mean values of the PET-derived functional primary endpoints (Volume of distribution, and/or some form of integrated SUV) in this

population. Therefore our sample size is driven by a mixture of:

- (i) what is known about between-subject variability from relevant, recent PET studies,
- (ii) feasibility, and
- (iii) flexibility.

An ongoing study investigating the validation and dosimetry of a PET ligand in healthy subjects and patients with IPF (study RES116235) has been able to draw firm conclusions about similar endpoints (in terms of the estimation methods we describe below) using around 5 subjects. Therefore we will set five patients and five age-matched HVs as our initial target sample size.

From that point onwards, the data will be monitored continuously (or as near as possible given practicalities of study operationalisation), and at each step the following decisions will be made:

- Stop, and conclude that there is strong evidence of differential FAK expression (as measured by the study endpoints) between patients and HVs.
- Stop, and conclude that there is insufficient evidence of any great difference, and furthermore (conditional on observed data i.e. in a formal Bayesian sense) there is low probability that an increase in sample size will reverse such a conclusion
- Continue to enrol patient-HV pairs, and re-evaluate the decision.

This iterative cycle will be followed up until a maximum of twelve patients and twelve HVs have been recruited into the study.

## 8.1 Sample Size Re-estimation or Adjustment

The first statistical evaluation of the data will occur once five patients and five healthy volunteers have been studied in the PET scanner, and the relevant functional endpoints (such as  $V_T$ ) have been derived from their scan data by Imanova scientists. At this point, the statistical analysis (set out below) will be carried out, and, based on those results, the team may decide to recruit more subjects, up to a total of twelve patients and twelve healthy volunteers.

## 9 Analysis Populations

The following populations will be identified:

Screened Population: all subjects who signed an informed consent form and were

evaluated for study participation.

Safety Population: All patients and subjects who received the microdose of

study drug.

The primary endpoint will be analysed using the Safety Population.

### 9.1 Analysis Datasets

All analysis datasets will be based on observed data, except as outlined in Section 12.2.

## 10 Treatment Comparisons

The comparison of interest is uptake of [11C]-GSK2256098 in PAH patients versus healthy volunteers.

## 11 General Considerations for Data Analyses

## 11.1 Data Display Group Descriptors

The sort order for groups will be PAH patients then healthy control subjects. When a total column is included, it immediately follows the groups which it aggregates.

Listings of data will be sorted and displayed by group, subject number, and also by date and time if applicable.

The group descriptions to be used on all tables and listings are:

#### **Groups**

PAH Patients Healthy Volunteers

### 11.2 Conventions for Summary Statistics and Data Displays

The minimum set of summary statistics for numeric variables will be: n, mean, standard deviation (or standard error), median, minimum and maximum

Categorical data will be summarised in frequency tables with n and percentage. Summaries of a categorical variable will include all recorded values.

The minimum and maximum values will be presented with the same number of decimal places as the raw data collected on the CRF (or to 3 significant figures for derived parameters). The mean and percentiles (e.g. median, Q1, and Q3) will be presented using one additional decimal place. The standard deviation and standard error will be presented using two additional decimal places.

## 12 Data Handling Conventions

### 12.1 Premature Withdrawal and Missing Data

All subjects who withdraw prematurely from the study or study drug will be included in the statistical analyses.

If a subject completes the treatment period but has missing data, then this will be made apparent in the subject listings. Missing data will not be imputed except for as outlined in Section 12.2.

If the study is prematurely discontinued, all available data will be listed and a review will be carried out to assess which statistical analyses are still considered appropriate.

Data collected at unscheduled time points during the study will not be used in the summaries or data analyses. They will be included in the listings.

If time information (i.e. hours and/or minutes) for adverse events or concomitant medication is missing, but the day is present, then the time will be calculated in days. If date information is partial or missing, then any derived times (e.g. AE start time from last study medication) will be listed as missing.

#### 12.2 Derived and Transformed Data

 $V_T$  and mean SUV will be derived by Imanova for regions including heart chamber and whole lung.

The CT images obtained for attenuation correction (AC) of the PET [CT-AC)] are used to delineate the left and right lung and both the CT-AC and the region of interest (ROI) image are resampled to the PET space. Time activity curves are extracted using the predefined ROI image. Standardized uptake values (SUV) are generated by averaging the time activity curves between two time points (to be defined depending on the kinetics of the tracer in the lungs) and normalising to the injected dose per unit mass.

An image derived input function is generated using a region of interest in the pulmonary artery. This input function is used together with a compartmental model to derive the volume of distribution  $(V_T)$  in each region of interest.

#### 12.3 Assessment Windows

No assessment windows are defined for this report.

#### 12.4 Values of Potential Clinical Importance

Any laboratory value outside the reference range for that variable (Appendix B) will be flagged as a value of a potential clinical importance

A vital signs result will be considered to be of potential clinical importance if it falls outside the relevant range below:

| Vital Sign | Range |
|------------------------------------------------|------------------|
| Supine/semi-recumbent systolic blood pressure | 85–160 mm Hg |
| Supine/semi-recumbent diastolic blood pressure | 40–90 mm Hg |
| Supine/semi-recumbent heart rate | 40–100 beats/min |
| Respiration rate | 8–20 per min |
| Oral temperature | 35.5–37.8°C |

## 13 Study Population

## 13.1 Disposition of Subjects

All analyses will use the safety population.

The disposition of all subjects (patients and healthy volunteers) in the safety population will be summarised including number of subjects screened, the number of subjects who failed screening, number completing the study by group, and number withdrawn from the study.

All subjects who withdraw or are withdrawn from the study will be listed by treatment, with the reason for withdrawal.

A listing of analysis populations will be provided.

#### 13.2 Protocol Deviations

Before closing the database, data listings will be reviewed to identify any significant deviations and determine whether the data should be excluded from any analysis populations.

Major protocol deviations include subjects who:

- Entered the study even though they did not satisfy the entry criteria.
- Met the criteria for withdrawal from the study but were not withdrawn.
- Received the wrong treatment or incorrect dose.
- Received an excluded concomitant therapy.
- Received investigational product(s) past the expiration date.
- Healthy volunteers who are not matched to a PAH patient on gender or with age not within  $\pm$  5 years

A summary table of the important deviations will be provided.

A listing of inclusions/ exclusion deviations will be provided.

A listing of all important deviations will be provided.

## 13.3 Demographic and Baseline Characteristics

Demographic and baseline characteristics (e.g. physical examination, vital signs, Allen's test and INR) will be listed and summarised. A summary of age ranges of subjects will be presented.

A summary of the difference in ages between the matched pairs will also be presented.

Subjects who take concomitant medication will be listed. All non-trial medication will be coded by GSK.

### 13.4 Treatment Compliance

Dates and times of dosing will be listed (Listing 16.2.1.1).

## 14 Safety Analyses

The dates and times of treatment dosing will be listed to indicate exposure to the study medication (Listing 16.2.1.1).

#### 14.1 Adverse Events

Adverse events will be coded by GSK.

All adverse events will be listed. Subject numbers for specified adverse events will be listed. A listing of the relationship between system organ class and verbatim text will also be presented.

The number of subjects with at least one treatment-emergent adverse event (TEAE) will be tabulated by actual treatment and MedDRA system organ class. A treatment-emergent adverse event is defined as an event emerging during treatment having been absent pretreatment or having worsened relative to pre-treatment<sup>1</sup>.

For each of the following, the number of subjects with adverse events will be summarised:

- TEAEs by system organ class and preferred term
- IMP-related (as recorded by the Investigator) TEAEs by system organ class and preferred term

Subjects with more than one TEAE will be counted only once, at causality, for each system organ class/preferred term. Multiple TEAEs in a subject will be counted once per system organ class and preferred term. Adverse events with missing severity and/or causality will be treated as severe and related to IMP, respectively.

Summaries will be sorted by system organ class and decreasing total incidence of preferred term.

#### 14.2 Serious Adverse Events

Serious Adverse Events will be summarised by by system organ class and preferred term.

A listing of the reasons for considering a serious adverse event will be provided.

### 14.3 Other Safety Measures

#### 14.3.1 Clinical Laboratory Evaluations

All laboratory values of potential clinical importance will be listed.

#### 14.3.2 Vital signs

Vital signs evaluation pre- and post-scan at the scanning visit will be summarised by group. Vital signs of potential clinical importance will be listed.

#### 14.3.3 Physical examination

Abnormal physical examination findings will be listed by group.

#### 14.4 Positron Emission Tomography

Positron Emission Tomography (PET) parameters will be summarised using the safety population.

Each PET parameter (V<sub>T</sub> and mean SUV) will be listed and summarised by region and group.

A Bayesian approach to the analysis of the PET parameters will be used.

For any important endpoint, we describe our uncertainty concerning its true value with a probability density function,  $p(\theta)$ , say. (Suppose ' $\theta$ ' represents Volume of Distribution, derived from the PET and blood sample data. The following argument will apply to any such endpoint which takes numerical values on the real line.) Pre-study start, we will characterise  $p(\theta)$  in such a way that our "prior belief" about the true endpoint's value is entirely diffuse over the real line (this approach implies that all conclusions about the endpoint are driven only by the data gathered in the study).

We will gather evidence about the endpoint in the data from the study, which we will characterise via its likelihood function (derived from the relevant sampling distribution,  $l(x|\theta)$ , say, where 'x' stands for 'data'). From the likelihood function the usual summary statistics for the endpoint are derived.

It is highly likely, based on similar PET studies, that a Normal likelihood function will be suitable. This will have an unknown mean and known variance taken from the raw data (i.e.

 $x_j \sim N(\theta_j, \sigma_j^2)$  where j is the PAH patient group or the HV group). An uninformative conjugate Normal prior density function with mean zero and a vast variance will be adopted for the group mean  $(P(\theta_j) = N(0, \sigma_{0,j}^2))$  leading to the standard Normal posterior density functions for the endpoints of interest (Should the data not support a Normal likelihood function, alternative parametric forms, such as a log-Normal density, will be investigated). In order for the prior to be sufficiently non-informative, the variance of the prior will be approximately 100 times the variance of the data.

We will apply Bayes' theorem to derive the posterior density function  $p(\theta_j \mid x_j)$ . We will use PROC MCMC in SAS. The number of burn-in iterations will be at least 10,000 and the number of MCMC iterations, excluding the burn-in iterations will be at least 5000. These samples may be thinned if autocorrelation is high. An example of the SAS code for a normal likelihood function is given below:

```
ods output PostSummaries = PostSummaries PostIntervals = PostIntervals
PosteriorSample = PosteriorSample;
```

```
PROC MCMC data = BayesianTest nmc = 5000 nbi = 10000 monitor=(_parms_ muratio);

parms mu1 mu2;

muratio = mu1/mu2;

MODEL PAH ~ norm(mu1, sd = 1;

MODEL HVs ~ norm(mu2, sd = 1);

prior mu1 mu2 ~ normal(0, sd = 100);

preddist outpred = BayesianPred nsim = 5000 covariates = PredCovariates;

by endpoint region;

run;
```

The posterior distribution for each endpoint will be summarised by region and group, including the mean, median, SD, interquartile range and 95% credible interval based on the highest posterior density (HPD) interval.

Samples from the posterior distribution for the group mean  $p(\theta_j|x_j)$  for the PAH patients and for the HV subjects will be used to determine the posterior distribution for the ratio of group means (PAH patients to HV subjects). The posterior distribution for the ratio of group means

will be summarised by region and endpoint. Plots of the median and 95% credible interval for the posterior distribution of the group mean and the ratio of group means will be presented for each endpoint and region. Individual subject data will also be included on the plot using a different symbol for each match pairs of subjects. Each plot will also include the posterior distribution of the ratio of the group means.

Samples from the posterior distribution of the ratio of group means will be used to determine the probability that the ratio of the endpoint in PAH patients to HV subjects exceeds 1 for each endpoint and region. This will be repeated for other values to allow us to plot to provide a graph of the "probability that this ratio exceeds a certain value, plotted against ratio, for ratios in the range 0.5 to 2 will be presented for each endpoint and region.

#### 15 References

- 1. International Conference on Harmonization, 1998. Statistical Principles for Clinical Trials ICH Harmonised Tripartite Guideline. Guidance for Industry, E9, FDA federal register, Vol 63, 1998, p49583. Available at: http://www.fda.gov/cder/guidance.
- 2. International Conference on Harmonization, 1995. Structure and Content of Clinical Study Reports ICH Harmonised Tripartite Guideline. Guidance for Industry, E3, FDA federal register, Vol 61, 1996, p37320. Available at: http://www.fda.gov/cder/guidance.

#### 16 ATTACHMENTS

#### 16.1 Data Display Requirements

Data displays will be stored in individual PDF files with formatting of:

- pagesize will be 8.5" x 11" (US Letter sized paper)
- margins will be 1.25" top and bottom and 0.87" right and left on a landscape page
- font will be Arial 10.

There will be a bookmark to the first page of each display. Bookmark text will include display type (Table, Figure, Listing), display number and the verbatim text of the data display. Bookmarks will link directly to the first page of the data display rather than executing a Java script.

## 16.2 Table of Contents for Data Display Specifications

For overall page layout refer to Appendix A.

The numbering in the tables below will take precedence over the numbering in the shells.

The following tables and figures will be produced (templates provided in Section 16.2 and 16.3):

The following tables and figures will be produced (templates provided in Section 16.2.1 and 16.2.2):

| Table | Description | Population | Source<br>Listing | Template (Shells below) |
|---|---|---|---|---|
| 10.1 | Summary of Subject Disposition | Screened | 16.2.1.2,<br>16.2.3.1 | T SD1 |
| 10.2 | Summary of Important Protocol Deviations | Safety | 16.2.2.2 | T DV GK |
| 14.1 | DEMOGRAPHIC DATA | | | |
| 14.1 | Summary of Demographic Characteristics | Safety | 16.2.4.1 | T DM1 PG |
| 14.2 | Summary of Age Ranges | Safety | 16.2.4.1 | T AGE GSK |
| 14.3 | Summary of Age Matching | Safety | 16.2.4.1 | <u>T_DM2</u> |
| 14.3 | SAFETY DATA | | | |
| 14.3.1.1 | Summary of Treatment-Emergent Adverse Events | Safety | 16.2.7.1 | T AE1 |
| 14.3.1.2 | Summary of Drug-Related Treatment-Emergent Adverse Events | Safety | 16.2.7.1 | <u>T AE1</u> |
| 14.3.2 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | Safety | 16.2.7.1 | T AE2 |
| 14.3.3 | Narratives of deaths and other serious adverse events | Safety | 16.2.7.1 | - |
| 14.3.4 | Summary of Vital Signs at Scanning Visit | Safety | - | <u>T VS1</u> |
| 14.4 | PET DATA | | | _ |
| 14.4.1 | Summary of Volume of Distribution $(V_T)$ and Mean Standardised Uptake Values (SUV), by Group and Region | Safety | 16.2.9.1 | T PT1 GK |
| 14.4.2 | Summary of the Posterior Distribution for Volume of Distribution $(V_T)$ and Mean Standardised Uptake Values (SUV), by Group and Region | Safety | 16.2.9.1 | T_PT2_GK |
| 14.4.3 | Summary of the Posterior Distribution of the Ratio of Group Means for Volume of Distribution (V <sub>T</sub> ) and Mean Standardised Uptake Values (SUV), by Region | Safety | 16.2.9.1 | T PT3 GK |
| 14.4.4 | Posterior Probability that the Ratio of Group Means for Volume of Distribution $(V_T)$ and Mean Standardised Uptake Values (SUV) Exceeds a Certain Value, by Region | Safety | 16.2.9.1 | T PT4 GK |

| Figure | Description | Population | Source<br>Listing | Template (Shells below) |
|---|---|---|---|---|
| 14.1 | PET DATA | Safety | | |
| 14.1.1.1 | Plot of the Posterior Distribution of the Volume of Distribution (V <sub>T</sub> ) for<br>the Group Means and the Ratio of the Group Means, by Region | Safety | 16.2.9.1 | F PT1 GK |
| 14.1.1.2 | Plot of the Posterior Distribution of the Mean Standardised Uptake<br>Values (SUV) for the Group Means and the Ratio of the Group Means,<br>by Region | Safety | 16.2.9.1 | F PT1 GK |
| 14.1.2.1 | Plot of the Posterior Probability that the Ratio of the Group Means Exceeds a Certain Value for the Volume of Distribution $(V_T)$ , by Region | Safety | 16.2.9.1 | F PT2 GK |
| 14.1.2.2 | Plot of the Posterior Probability that the Ratio of Group Means Exceeds<br>a Certain Value for Mean Standardised Uptake Values (SUV), by<br>Region | Safety | 16.2.9.1 | F_PT2_GK |

The following abbreviated listings will be produced (templates provided in Section 16.2.3):

| Listing | Description | Template (Shells below) |
|---|---|---|
| 16.2.1 | Study dates & disposition of subjects | |
| 16.2.1.1 | Listing of Study Dates | L SD1 PG |
| 16.2.1.2 | Listing of Reasons for Withdrawal | L SD2 PG |
| 16.2.2 | Protocol deviations | |
| 16.2.2.1 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | L DV1 PG |
| 16.2.2.2 | Listing of Important Protocol Deviations | L DV2 PG |
| 16.2.3 | Analysis sets, including subjects excluded from analysis | |
| 16.2.3.1 | Listing of Analysis Populations | L AN1 PG |
| 16.2.4 | Demographic data & concomitant medication | |
| 16.2.4.1 | Listing of Demographic Characteristics | L DM1 PG |
| 16.2.4.2 | Listing of Concomitant Medications | L CM1 PG |
| 16.2.5 | Study drug administration | |
| 16.2.5.1 | Listing of Exposure Data | L EX1 PG |

| 16.2.7 | Adverse events | |
|---|---|---|
| 16.2.7.1 | Listing of All Adverse Events | L AE1 PG |
| 16.2.7.2 | Listing of Serious Adverse Events | L AE1 PG |
| 16.2.7.3 | Listing of Adverse Events Leading to Withdrawal from Study | L AE1 PG |
| 16.2.7.4 | Listing of Subject Numbers for Specified Adverse Events | L AE1 GSK |
| 16.2.7.5 | Listing of Reasons for Considering a Serious Adverse Event | L AE3 GSK |
| 16.2.7.6 | Listing of Relationship between System Organ Class and Verbatim Text | L AE2 GSK |
| 16.2.8 | Laboratory values | |
| 16.2.8.1 | Listing of Clinical Chemistry Abnormalities of Potential Clinical | L LB1 PG |
| 10.2.6.1 | Importance | L LDI FU |
| 16.2.8.2 | Listing of Haematology Abnormalities of Potential Clinical Significance | <u>L LB1 PG</u> |
| 16.2.8 | Vital signs, ECGs and physical findings | |
| 16.2.8.1 | Listing of Vital Signs of Potential Clinical Importance | L VS1 PG |
| 16.2.8.2 | Listing of ECG data | L EG1 PG |
| 16.2.6.3 | Listing of Abnormal ECG Findings | L EG2 PG |
| 16.2.9 | PET Data | |
| 16.2.9.1 | Listing of Volume of Distribution (V <sub>T</sub> ) and Mean Standardised Uptake Values (SUV) | L PET GK |

## 16.3 Data Display Specifications

#### 16.3.1 Table Outlines

#### Template T\_SD1

Table 10.1 Summary of Subject Disposition

| | | | | Healthy | |
|---|---|---|---|---|---|
| Population | Status | Reason for Withdrawal | PAH Patients | Volunteers | All Subjects |
| Screened population | Included | | | | |
| | Failed screening | | | | |
| Safety population | Included | | | | |
| | Completed | | | | |
| | Withdrawn | | | | |
| | | Adverse Event | | | |
| | | Lack of efficacy | | | |
| | | Subject reached protocol- | | | |
| | | defined stopping criteria | | | |
| | | Study closed/terminated | | | |
| | | Lost to follow-up | | | |
| | | Investigator discretion | | | |
| | | Withdrew consent | | | |

Source: Listing 16.2.xx

Programming notes: Continued with all treatment groups.

#### Template T\_DV\_GK

Table 10.2 Summary of Important Protocol Deviations

| | PAH Patients | Healthy Volunteers |
|---|---|---|
| | (N=xx) | (N=xx) |
| Category/Subcategory | n (%) | n (%) |
| Any protocol deviations | 20 (20%) | 22 (22%) |
| Assessments and/or procedures | 10 (10%) | 8 (8%) |
| Failure to report SAE, pregnancy, or liver function abnormalities per protocol | 4 (4%) | 6 (6%) |
| Randomization procedures | 4 (4%) | 6 (6%) |
| Study treatment supply procedures | 4 (4%) | 6 (6%) |
| Other | 4 (4%) | 6 (6%) |
| Eligibility criteria not met | 6 (6%) | 8 (8%) |
| Not withdrawn after developing withdrawal criteria | 10 (10%) | 8 (8%) |
| Not discontinued from study treatment | 4 (4%) | 6 (6%) |
| Not withdrawn from study | 6 (6%) | 8 (8%) |
| Received wrong treatment or incorrect dose | 10 (10%) | 8 (8%) |
| Prohibited medication or device | 4 (4%) | 6 (6%) |
| Visit Window | 10 (10%) | 8 (8%) |
| Other protocol deviation category | 6 (6%) | 8 (8%) |

Source: Listing 16.2.xx

### Template T\_DM1

Table 14.1 Summary of Demographic Characteristics

| Variable | Statistics | PAH Patients<br>(N=xx) | Healthy Volunteers<br>(N=xx) | All Subjects<br>(N=xx) |
|---|---|---|---|---|
| Age (y) | n | (14-77) | (14-11) | (14-77) |
| 0 1,,, | Mean | | | |
| | SD | | | |
| | Min | | | |
| | Median | | | |
| | Max | | | |
| Gender | | | | |
| | Female (%) | | | |
| | Male (%) | | | |
| Race | American Indian or Alaskan | | | |
| | Native (%) | | | |
| | Asian (%) | | | |
| | Black (%) | | | |
| | Native Hawaiian or other | | | |
| | Pacific Islander (%) | | | |
| | White (%) | | | |
| | Other (%) | | | |
| Ethnicity | Hispanic or Latino (%) | | | |
| | Not Hispanic or Latino (%) | | | |
| Height (cm) | n | | | |
| | Mean | | | |
| | SD | | | |
| | Min | | | |
| | Median | | | |
| | Max | | | |
| Weight (kg) | n | | | |
| | Mean | | | |
| | SD | | | |
| | Min | | | |

| Variable | Statistics | PAH Patients<br>(N=xx) | Healthy Volunteers (N=xx) | All Subjects<br>(N=xx) |
|---|---|---|---|---|
| | Median | (IV-XX) | (11-22) | (11-22) |
| | Max | | | |
| BMI (kg/m2) | n | | | |
| | Mean | | | |
| | SD | | | |
| | Min | | | |
| | Median | | | |
| | Max | | | |
| Smoker | Yes (%) | | | |
| | No (%) | | | |
| Cigarettes* | n | | | |
| (Pack Years) | Mean | | | |
| | SD | | | |
| | Min | | | |
| | Median | | | |
| | Max | | | |
| Optional | | | | |
| (units) | | | | |

\*includes only those subjects who smoke Source: Listing 16.2.xx

Programming notes: Continued with all treatment groups and additional demographic characteristics

#### Template T\_AGE\_GSK

Table 14.3.6.xx Summary of Age Ranges

| | No Treatment | Treatment A | Treatment B | Total |
|---|---|---|---|---|
| | (N=1) | (N=100) | (N=100) | (N=201) |
| Age Ranges | | | | |
| In utero | 0 | 2 (2%) | 2 (2%) | 4 (2%) |
| Preterm newborn infants (gestational age <37 weeks) | 0 | 1 (1%) | 1 (1%) | 2 (1%) |
| Newborns (0-27 days) | 0 | 3 (3%) | 3 (3%) | 6 (3%) |
| Infants and toddlers (28 days-23 months) | 0 | 4 (4%) | 4 (4%) | 8 (4%) |
| Children (2-11 years) | 0 | 3 (3%) | 3 (3%) | 6 (3%) |
| Adolescents (12-17 years) | 0 | 1 (1%) | 1 (1%) | 2 (1%) |
| Adult (18-64 years) | 0 | 59 (59%) | 59 (59%) | 118 (59%) |
| >=65-84 years | 0 | 26 (26%) | 26 (26%) | 52 (26%) |
| >=85 years | 1 (100%) | 1 (1%) | 1 (1%) | 3 (1%) |

#### Template T\_DM2

Table 14.3.6.xx Summary of Age Matching

| | | Differer | nce in matched pai | rs (PAH-H) | /) |
|----|------|----------|--------------------|------------|-----|
| n* | Mean | SD | Median | Min | Max |

Source: Listing 16.2.xx

Programming notes: Add the footnote  $n^*$  number of matched pairs

#### Template T\_AE1

Table 14.3.3.xx Summary of Treatment-Emergent Adverse Events

| | | PAH Patie | nts (N=xx) | Healthy Volunteer<br>(N=xx) | |
|---|---|---|---|---|---|
| System Organ Class | Preferred Term | n | % | n | % |
| Number of subjects with AEs | | | | | |
| Gastrointestinal disorders | Total number of subjects | | | | |
| | Abdominal discomfort | | | | |
| | Abdominal pain | | | | |
| | <b>↓</b> | | | | |
| Nervous system disorders | Total number of subjects | | | | |
| | Dizziness | | | | |
| | Headache | | | | |
| | <b>↓</b> | | | | |
| <b>↓</b> | <b>↓</b> | | | | |

<sup>\*</sup>Subjects with ≥1 adverse event are counted only once per system organ class and preferred term.

Source: Listing 16.2.xx

Programming notes: Continued with all treatment groups

SOCs and PTs are sorted in decreasing order of frequency

Presented for all applicable MedDRA system organ classes and terms.

#### Template T\_AE2

Table 14.3.2x Summary of Serious Adverse Events by System Organ Class and Preferred Term

| System Organ Class<br>Preferred Term | | PAH Patients<br>(N=100) | Healthy Volunteers<br>(N=200) |
|---|---|---|---|
| ANY EVENT | Number of Subject with SAEs | 40 (40%) | 40 (20%) |
| | Number of SAEs | 50 | 50 |
| | Number of Drug-related SAEs | 20 | 20 |
| | Number of Fatal SAEs | 10 | 10 |
| | Number of Drug-related Fatal SAEs | 5 | 5 |
| Infections and infestations | | | |
| Diabetic Gangrene | Number of Subject with SAEs | 10 (10%) | 1 (<1%) |
| | Number of SAEs | 15 | 1 |
| | Number of Drug-related SAEs | 5 | 0 |
| | Number of Fatal SAEs | 2 | 0 |
| | Number of Drug-related Fatal SAEs | 1 | 0 |
| Erysipelas | Number of Subject with SAEs | 1 (<1%) | 10 (5%) |
| | Number of SAEs | 1 | 15 |
| | Number of Drug-related SAEs | 0 | 5 |
| | Number of Fatal SAEs | 0 | 2 |
| | Number of Drug-related Fatal SAEs | 0 | 1 |

#### Template T\_VS1

Table 14.3.6.xx Summary of Vital Signs at Scanning Visit

| | Group | Timepoint | n | Mean | SD | Median | Min | Max |
|---|---|---|---|---|---|---|---|---|
| Systolic BP (mmHg) | PAH Patients (N=xx) | | | | | | | |
| | Healthy Volunteers (N=xx) | | | | | | | |

Source: Listing 16.2.xx

Programming notes: Continued with all variables, treatments and time points

#### Template T\_PT1\_GK

Table 14.3.6.xx Summary of Volume of Distribution (V<sub>T</sub>) and Mean Standardised Uptake Values (SUV), by Group and Region

| Parameter (units) | Region | Group | n | Mean | SD | Median | Min | Max |
|---|---|---|---|---|---|---|---|---|
| Mean SUV | | PAH Patients (N=xx) | | | | | | |

Mean SUV is calculated over a xx minute period

Source: Listing 16.2.xx

Programming notes: Continued with all variables, groups and time points. Replace xx with the time period in the footnote.

#### Template T\_PT2\_GK

Table 14.3.6.xx Summary of the Posterior Distribution for Volume of Distribution (V<sub>T</sub>) and Mean Standardised Uptake Values (SUV), by Group and Region

| | | | | | Posterior distribution P(Θ /x) | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Parameter | Region | Group | Prior Distribution for Θ | Value of σ<br>used in then<br>model | Mean | SD | Median | 25th<br>quartile | 75th<br>quartile | 95% Credible Interval |
| Mean SUV | Heart Chamber | PAH Patients (N=xx) | normal(0, sd = 100) | 1 | | | | | | |
| | | Healthy Volunteers (N=xx) | normal(0, sd = 100) | 1 | | | | | | |
| | Whole Lung | | | | | | | | | |

Number of MCMC iterations, excluding the burn-in iterations = 5,000. Number of burn-in iterations = 10,000

The PET parameters are assumed to follow a normal distribution with unknown mean  $\Theta$  and known variance  $\sigma^2$  (i.e.  $N(\Theta, \sigma^2)$ )

 $P(\Theta|X)$  is the posterior distribution for  $\Theta$  given the PET data x. 95% credible intervals based on the highest posterior density interval.

Mean SUV is calculated over a xx minute period

Source: Listing 16.2.xx

Programming notes: Continued with all end points, regions and groups. Replace xx with the time period in the footnote.

#### Template T\_PT3\_GK

Table 14.4.3 Summary of the Posterior Distribution of the Ratio of Group Means for Volume of Distribution (V<sub>T</sub>)and Mean Standardised Uptake Values (SUV), by Region

| | | Posterior Distribution $P(\Theta_{PAH} x_{PAH})/P(\Theta_{HV} x_{HV})$ | | | | | |
|---|---|---|---|---|---|---|---|
| variable | Region | Mean | SD | Median | Min | Max | 95% Credible Interval |
| Mean SUV | Heart Chamber | | | | | | |
| | Whole Lung | | | | | | |

Number of MCMC iterations, excluding the burn-in iterations = 5,000. Number of burn-in iterations = 10,000 95% credible intervals based on the highest posterior density interval.

Note: PAH = PAH Patients, HV = Healthy Volunteers

Source: Listing 16.2.xx

#### Template T\_PT4\_GK

Table 14.3.6.xx Posterior Probability that the Ratio of Group Means for Volume of Distribution (V<sub>T</sub>) and Mean Standardised Uptake Values (SUV) Exceeds a Certain Value, by Region

| Mean SUV |
|----------|

Note: P(ratio) > 1 is the probability that the posterior ratio of group means exceeds 1 based on 5,000 simulated posterior predicted values

\*Ratio of PAH patients to Healthy Volunteers.\*

\*Mean SUV is calculated over a xx minute period\*

Source: Listing 16.2.xx

Programming notes: Continued with all variables. Replace xx with the time period in the footnote.

## 16.3.2 Figure Outlines

#### Template F\_PT1\_GK

Figure 14.3.6.xx Plot of the Posterior Distribution of the Volume of Distribution (V<sub>T</sub>) for the Group Means and the Ratio of the Group Means, by Region



95% credible intervals based on the highest posterior density interval. Programming note: use the same symbols for each of the matched pairs

#### Template F\_PT2\_GK

Figure 14.3.6.xx Plot of the Posterior Probability that the Ratio of the Group Means Exceeds a Certain Value for the Volume of Distribution (V<sub>T</sub>), by Region



### 16.3.3 Listing Outlines

Template L\_SD1\_PG

Listing 16.2.x.xx Listing of Study Dates

Group Subject Screening Scanning visit Follow Up

Template L\_SD2\_PG

Listing 16.2.x.xx Listing of Reasons for Withdrawal

Date of Study

Group Subject Withdrawal Day Reason

Template L\_DV1\_PG

Listing 16.2.x.xx Listing of Subjects with Inclusion/Exclusion Criteria Deviations

Group Subject Type Criterion

Inclusion

Exclusion

Template L\_DV2\_PG

Listing 16.2.2.3 Listing of Subjects with Important Protocol Deviations

Group Subject Protocol Deviation

Template L\_AN1\_PG

Listing 16.2.x.xx Listing of Analysis Populations

Group Subject Population Population

#### Template L\_DM1\_PG

Listing 16.2.x.xx Listing of Demographic Characteristics

| Group | Subject | Date of visit | Year of<br>birth | Age (y) | Gender | Race | Ethnicity | Height (c | m) Weight ( | kg) BMI (kg/m2 |
|---|---|---|---|---|---|---|---|---|---|---|
| PAH Patients | | | | | | | | | | |
| Healthy | | | | | | | | | | |
| Volunteers | | | | | | | | | | |
| Group | Subject | Smoking | Da | ite Last | Cigarettes | Number | r Years | Cigarettes | Allen's Test | INR (units) |
| | | Status | Sn | noked | (daily) | Smoked | ł | (Pack Years) | | |
| PAH Patients | | | | | | | | | | |
| Healthy | | | | | | | | | | |
| Volunteers | | | | | | | | | | |

#### Template L\_CM1\_PG

Listing 16.2.x.xx Listing of Concomitant Medications

| | | | Dose/ | | | | |
|---|---|---|---|---|---|---|---|
| | | Drug Name/ | Units/ Freq/ | Date/time Started/ | Time Since Last | Started Pre- | Ongoing |
| Group | Subject | Indication | Route | Date Stopped | Dose | Trial? | Medication? |

#### Template L\_EX1\_PG

Listing 16.2.x.xx Listing of Exposure Data

| | | | | Dur- | | | | |
|---|---|---|---|---|---|---|---|---|
| | | Start Date/ | Stop Date/ | ation | | Dose | Formulation/ | • |
| Group | Subject | Start Time of Dose | Stop Time of Dose | (days) | Dose | Unit | Route | Frequency |
| PAH Patients | PPD | PPD | PPD | 46 | 25 | mg | Tablet/ | 2xday |
| | | | | | | | Oral | |

#### Template L\_AE1\_PG

Listing 16.2.x.xx Listing of All Adverse Events

| | | | | | | | Frequency/ Action | Related to Study |
|---|---|---|---|---|---|---|---|---|
| | | System Organ Class/ | Outcome/ | Onset ( | | Severity/ | Taken (1)/ | Treatment/ |
| | | Preferred Term/ | Date/Time/ Resolved | | Time Since Last | Serious/ | Other Action | Treatment |
| Group | Subject | Verbatim Text | Date/Time | e/ Duration | Dose | Withdrawal | Taken | Emergent? |
| PAH Patients | PPD | Gastrointestinal disorders / | Resolved/ | | 10d 7h 3m | Mild/ | Intermittent/ Dose | Possibly/ |
| | | Intestinal spasm/ | PPD | 13:05/ | | No/ | not changed/ | Yes |
| | | Entero-spasm | PPD | 7:50/ | | Yes | None | |
| | | | 34d 4h 5m | 1 | | | | |

<sup>(1)</sup> Action Taken with Study Treatment

Template L\_AE1\_GSK

#### 16.2.7.4 Listing of Subject Numbers for Specified Adverse Events

| System Organ Class/<br>Preferred Term | Group | No.<br>with<br>Event | Unique Subject Id. |
|---|---|---|---|
| Gastrointestinal disorders/<br>Dyspepsia | PAH Patients | x | PPD |

Template L\_AE2\_GSK

#### 16.2.7.6 Listing of Relationship between System Organ Class and Verbatim Text

| System Organ Class | Preferred Term | Verbatim Text |
|---|---|---|
| Blood and lymphatic system disorders | Lymphadenopathy | ENLARGED LYMPH NODE |
| Cardiac disorders | Palpitations<br>Tachycardia nos | HEART PALPITATION TACHYCARDIA |

#### Template L\_AE3\_GSK

#### 16.2.7.5 Listing of Reasons for Considering a Serious Adverse Event



- [1] Resulted in death.
- [2] Was life-threatening.
- [3] Required hospitalization or prolongation of existing hospitalization.
- [4] Resulted in persistent or significant disability/incapacity.
- [5] Congenital anomaly/birth defect.
- [6] Other medically important serious event.
- [7] Protocol specified serious event.

#### Template L\_LB1\_PG

Listing 16.2.x.xx Listing of Clinical Chemistry Abnormalities of Potential Clinical Importance

| | | | Planned | | | | |
|---|---|---|---|---|---|---|---|
| | | | Relative | | | | |
| Group | Subject | Lab test (units) | Time | Date/Time | Value | Range | NR |
| | PPD | Alk Phos (U/L) | | | | | L |
| | | | | | | | Н |
| | | ALT (U/L) | | | | | |

NR = Normal Range flag
H = Above reference interval, L = Below reference interval,

#### Template L\_VS1\_PG

Listing 16.2.x.xx Listing of Vital Signs of Potential Clinical Importance

| | | | | Systolic | Diastolic | |
|---|---|---|---|---|---|---|
| | | Planned Relative | | <b>Blood Pressure</b> | <b>Blood Pressure</b> | Etc |
| Group | Subject | Time | Date/Time | (mmHg) | (mmHg) | (units) |
| PAH Patients | | 24 H | 26SEP2012:09:57 | 63 | 148 <sup>*</sup> | |

<sup>\*</sup> Value of potential clinical importance

Template L\_EG1\_PG

Listing 16.2.x.xx Listing of ECG Values

| | | | | Heart | | QRS | QRS | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | Planned | | Rate | PR Int. | Dur. | Axis | QT int | QTcB | QTcF |
| Treatment | Subject | Relative Time | Date/Time | (bpm) | (msec) | (msec) | (deg) | (msec) | (msec) | (msec) |

Programming notes:

Template L\_EG2\_PG

Listing 16.2.x.xx Listing of Abnormal ECG Findings

| | | | Comment on Clinical | | |
|---|---|---|---|---|---|
| Treatment | Subject | Time | Date/Time | ECG Finding | Significance |

Programming notes: Lists only values with Normal variant='No' or with comment on ECG result

ECG Finding contains Physician's Opinion from CRF and relates to whole trace (not individual parameters), e.g. Normal, Abnormal - NCS or Abnormal - CS

#### Template L\_PE1\_PG

Listing 16.2.x.xx Listing of Abnormal Physical Examination Findings

Planned Relative

Group Subject Time Date/Time Site Details

Programming Notes: List only findings with an 'abnormal' result.

If subjects have multiple abnormal sites at a given time, create a separate row for each site.

#### Template L\_PET\_GK

Listing 16.2.x.xx Listing of Volume of Distribution ( $V_T$ ) and Mean Standardised Uptake Values (SUV)

Date/Start Time / Mean Standardised Volume of Distribution (V<sub>T</sub>)

Group Subject Stop Time Region Uptake Value (SUV) (mL/cm³)

Programming Notes: Add the footnote Mean SUV is calculated over a xx minute period. Note xx in the footnote will be replaced by the time period

# **Appendix A: Laboratory Ranges**

| Laboratory Assessments Parameters | | | | | Range for potential clinical concern | |
|---|---|---|---|---|---|---|
| | Unit | Sex | Max age | Normal Range | Low | High |
| Haematology | | | | | | |
| Platelet Count | 10^9/L | F | NA | 163 - 376 | 100 | 600 |
| Platelet Count | 10^9/L | M | NA | 129-346 | 100 | 600 |
| Red blood cell count | 10^12/L | F | NA | 3.7-5.1 | NA | NA |
| Red blood cell count | 10^12/L | M | NA | 4.4-6.0 | NA | NA |
| Neutrophils | 10^9/L | Both | NA | 1.57-6.81 | 1.2 | 13 |
| Hemoglobin | pg | F | NA | 114-153 | 110 | 175 |
| Hemoglobin | pg | M | NA | 133-170 | 125 | 185 |
| Lymphocytes | 10^9/L | Both | NA | 0.89-2.88 | 0.5 | 4 |
| Hematocrit | L/L | F | NA | 0.338-0.445 | 0.3 | 0.55 |
| Hematocrit | L/L | M | NA | 0.386-0.489 | 0.35 | 0.65 |
| MCV | | | | | NA | NA |
| MCH | | | | | NA | NA |
| MCHC | | | | | NA | NA |
| Monocytes | 10^9/L | Both | NA | 0.09-0.90 | NA | NA |
| Eosinophils | 10^9/L | Both | NA | 0.05-0.55 | NA | 0.55 |
| Basophils | 10^9/L | Both | NA | 0.00-0.14 | NA | NA |
| Cinical Chemistry | | | | | | |
| BUN (Urea) | mmol /L | F | 54 | 2.2- 6.7 | NA | 12 |
| BUN (Urea) | mmol /L | F | 120 | 3.0-8.6 | NA | 12 |
| BUN (Urea) | mmol /L | M | 54 | 2.7-7.6 | NA | 12 |
| BUN (Urea) | mmol /L | M | 120 | 3.0-8.6 | NA | 12 |
| Potassium | mmol/L | Both | NA | 3.5-5.3 | 3 | 5.5 |
| AST (SGOT) | lU/L | F | NA | <=30 | NA | 200 |
| AST (SGOT) | lU/L | M | NA | <=62 | NA | 200 |
| Total bilirubin | | F | NA | <= 19.7 | NA | 40 |
| Total bilirubin | | M | NA | <=29.3 | NA | 40 |
| Direct Bilirubin | | F | NA | <=3.9 | NA | NA |
| Direct Bilirubin | | M | NA | <=6.2 | NA | NA |
| Creatinine | | F | NA | 42-72 | NA | 150 |
| Creatinine | | M | NA | 53-102 | NA | 150 |
| Sodium | mmol/L | Both | NA | 133-146 | 125 | 160 |
| ALT (SGPT) | lU/L | F | NA | <=33 | NA | 200 |
| ALT (SGPT) | lU/L | M | NA | <=70 | NA | 200 |

| Total Protein | g/L | Both | NA | 60-80 | NA | NA |
|---------------|--------|------|----|---------|----|-----|
| Glucose | mmol/L | Both | NA | 2.8-5.8 | 2 | 10 |
| Calcium | mmol/L | Both | NA | 2.2-2.6 | 2 | 2.6 |
| Albumin | g/L | Both | NA | 35-50 | 30 | 60 |

## **Appendix B: Sample Page Layout**

| GlaxoSmithKline Ltd: 204746 | | |
|---|---|---|
| Population: [Pop] | | |
| | Table [number] [title] | |
| | Column headers | |
| | Main body of output | |
| | Source:Listing[16.2.xx] | |
| Footnotes about the table or listi | ing text go here. | |
| Program: [Prog Name] | [Date] | <br>HMR 15-505 |
| Produced By:[Username] | [Edito] | 7 IWIN 10 000 |
| *y = last page of individu | ual output | |